CLINICAL TRIAL: NCT00635024
Title: A Phase II Trial of Thymoglobulin and Melphalan in Patients With Relapsed Multiple Myeloma
Brief Title: Anti-thymocyte Globulin and Melphalan in Treating Patients With Relapsed Multiple Myeloma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Due to competing trials, this study is permanenlty closed to patient acrrual.
Sponsor: Mayo Clinic (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000589032; P30CA015083 (NIH); MC0687 (Other: Mayo Clinic Cancer Center); 06-005792 (Other: Mayo Clinic IRB)
Record Dates: First submitted 2008-03-12; First posted 2008-03-13 (Estimated); Results first posted 2010-10-18 (Estimated); Last update posted 2017-02-10 (Actual); Status verified 2011-08

CONDITIONS: Multiple Myeloma and Plasma Cell Neoplasm
Keywords: refractory multiple myeloma; stage I multiple myeloma; stage II multiple myeloma; stage III multiple myeloma
MeSH Terms: conditions — Multiple Myeloma; Neoplasms, Plasma Cell | interventions — Antilymphocyte Serum; Melphalan

ARMS (1):
- Anti-thymocyte Globulin/Melphalan (Experimental): Anti-thymocyte Globulin (2.5 mg/Kg)and Melphalan (16 mg/m^2)
  Interventions: Biological: anti-thymocyte globulin; Drug: melphalan

INTERVENTIONS:
Biological: anti-thymocyte globulin — 2.5 mg/kg
Drug: melphalan — 16 mg/m^2

SUMMARY:
RATIONALE: Biological therapies, such as anti-thymocyte globulin, may stimulate the immune system in different ways and stop cancer cells from growing. Drugs used in chemotherapy, such as melphalan, work in different ways to stop the growth of cancer cells, either by killing the cells or by stopping them from dividing. Anti-thymocyte globulin may also make cancer cells more sensitive to melphalan. Giving anti-thymocyte globulin together with melphalan may kill more cancer cells.

PURPOSE: This phase II trial is studying how well giving anti-thymocyte globulin together with melphalan works in treating patients with relapsed multiple myeloma.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To evaluate the hematological response rate of anti-thymocyte globulin given in combination with melphalan in patients with relapsed multiple myeloma.

Secondary

* To assess the toxicity and tolerability of this combination in these patients.
* To assess time to disease progression in patients treated with these drugs.
* To assess survival of patients treated with these drugs. OUTLINE: Patients receive anti-thymocyte globulin IV over 6 hours and melphalan IV on day 1. Treatment repeats every 28 days for 6 courses. Patients then receive melphalan alone as above for another 6 courses. Treatment continues in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed every 3 months until disease progression and then every 6 months for up to 2 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of multiple myeloma

  - Relapsed disease
* Must not be a candidate for stem cell transplantation, has refused transplantation, or has had stem cells collected previously
* Measurable disease, defined by ≥ 1 of the following:

  * Serum monoclonal protein ≥ 1.0 g by protein electrophoresis
  * More than 200 mg of monoclonal protein in the urine on 24 hour electrophoresis
  * Serum immunoglobulin free light chain ≥ 10 mg/dL AND abnormal serum immunoglobulin kappa to lambda free light chain ratio
  * Monoclonal bone marrow plasmacytosis ≥ 30% (evaluable disease)

PATIENT CHARACTERISTICS:

* Eastern Cooperative Oncology Group (ECOG) performance status 0-3
* Absolute neutrophil count ≥ 1,000/μL
* Platelet count ≥ 75,000/μL
* Hemoglobin ≥ 8.0 g/dL
* CD4 > 100/μL
* Creatinine ≤ 3 mg/dL
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No active malignancy with the exception of nonmelanoma skin cancer or in situ cervical or breast cancer
* No uncontrolled infection
* No other co-morbidity that would interfere with patient's ability to participate in trial

PRIOR CONCURRENT THERAPY:

* No limit to prior therapy
* At least 4 weeks since prior melphalan or other myelosuppressive agents
* At least 2 weeks since prior non-myelosuppressive agents (e.g., thalidomide or high-dose corticosteroids)
* No concurrent high-dose corticosteroids

  * Concurrent chronic steroids (maximum dose 20 mg/day prednisone equivalent) allowed if they are being given for disorders other than amyloid (e.g., adrenal insufficiency or rheumatoid arthritis)
  * Concurrent continuation of low level/stable steroid doses for replacement or inhalation therapy allowed
* Concurrent bisphosphonates allowed
* No concurrent immunosuppressive medications such as cyclosporine
* No other concurrent investigational treatment
* No concurrent cytotoxic chemotherapy or external-beam radiotherapy>
* No other concurrent systemic anti-neoplastic therapy including, but not limited to, immunotherapy, hormonal therapy, or monoclonal antibody therapy
* No concurrent prophylactic hematopoietic growth factors (unless for treatment of an established cytopenia)

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2008-05; Primary Completion 2008-07 (Actual); Study Completion 2010-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Shaji K. Kumar, MD, Study Chair — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: One (1) patient was recruited from May 2008 to September 2008 at Mayo Clinic. This trial was permanently closed in March 2009 due to competing trials.
Period: Overall Study
Arm/Group | Anti-thymocyte Globulin/Melphalan
Started | 1
Completed | 0
Not Completed | 1
Not completed — Adverse Event | 1

BASELINE CHARACTERISTICS:
Arm/Group | Anti-thymocyte Globulin/Melphalan
Number analyzed (Participants) | 1
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 1
  >=65 years | 0
Gender [Count of Participants; unit: Participants]
  Female | 1
  Male | 0
Region of Enrollment [Number; unit: participants]
  United States | 1
Prior Stem Cell Transplant [Number; unit: participants]
  Yes | 1
  No | 0
Parameters of Hematologic Response [Number; unit: participants] — Serum M-Spike >=1 g/dL
  participants
    Yes | 1
    No | 0
Parameters of Hematologic Response [Number; unit: participants] — Serum immunoglobulin free light chain >= 10 mg/dL
  participants
    Yes | 1
    No | 0
Parameters of Hematologic Response [Number; unit: participants] — Urine M-Spike >= 200 mg/24 hours
  participants
    Yes | 1
    No | 0
Parameters of Hematologic Response [Number; unit: participants] — Bone marrow plasma cells > 30%
  participants
    Yes | 1
    No | 0

OUTCOME MEASURES:

1. Primary Outcome: Hematological Response Rate Defined as the Number of Participants Who Achieve a Confirmed Response
Description: Response that was confirmed on 2 consecutive evaluations during the first 4 months of treatment.
  Complete Response(CR): Disappearance of M-protein from serum and urine, normalization of Free Light Chain (FLC) ratio and <5% plasma cells in bone marrow.
  Very Good Partial Response(VGPR): >=90% reduction in serum M-component; Urine M-Component <100mg per 24hours.
  Partial Response(PR): >=50% reduction in serum M-component and/or Urine M-Component >=90% reduction or <200mg per 24hours; or >=50% decrease in difference between involved and uninvolved FLC levels.
Time Frame: 4 months
Population: One participant was evaluable for the primary endpoint.
Measure: Number; unit: participants
Arm/Group | Anti-thymocyte Globulin/Melphalan
Number analyzed (Participants) | 1
participants | 0

2. Secondary Outcome: Overall Survival (OS)
Description: OS was defined as the time from registration to death of any cause.
Time Frame: up to 2 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Anti-thymocyte Globulin/Melphalan
Number analyzed (Participants) | 1
months | 2.9

3. Secondary Outcome: Progression-free Survival (PFS)
Description: PFS was defined as the time from registration to progression or death due to any cause.
  Progression was defined as any one or more of the following:
  An increase of 25% from lowest confirmed response in:
  * Serum M-component (absolute increase >= 0.5g/dl)
  * Urine M-component (absolute increase >= 200mg/24hour
  * Difference between involved and uninvolved Free Light Chain levels (absolute increase >= 10mg/dl)
  * Bone marrow plasma cell percentage (absolute increase of >=10%)
  * Definite development of new bone lesion or soft tissue plasmacytomas
Time Frame: up to 2 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Anti-thymocyte Globulin/Melphalan
Number analyzed (Participants) | 1
months | 2.9

4. Secondary Outcome: Duration of Response (DOR)
Description: DOR was calculated from the documentation of response (CR, VGPR or PR) until the date of progression in the subset of patients who responded.
Time Frame: up to 2 years
Population: All patients are non-evaluable - no patients responded to treatment.
Arm/Group | Anti-thymocyte Globulin/Melphalan
Number analyzed (Participants) | 0

5. Secondary Outcome: Number of Participants With Severe Non-hematological Adverse Events
Description: Severe non-hematologic adverse events were defined as adverse events grade 3 or higher, regardless of attribution to study drug. Adverse events were graded according to the National Cancer Institute Common Toxicity Criteria for Adverse Events (NCI CTCAE version 3.0)
Time Frame: every month during treatment, up to 12 months
Measure: Number; unit: participants
Arm/Group | Anti-thymocyte Globulin/Melphalan
Number analyzed (Participants) | 1
participants
  Yes | 1
  No | 0

ADVERSE EVENTS:
Arm/Group | Anti-thymocyte Globulin/Melphalan
Serious Adverse Events (participants affected / at risk) | 0/1
Other Adverse Events (participants affected / at risk) | 1/1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Anti-thymocyte Globulin/Melphalan (N=1)
Anemia (Blood and lymphatic system disorders) | 1 (1)
Hypersensitivity (Immune system disorders) | 1 (1)
Opportunistic Infection (Infections and infestations) | 1 (1)
Leukopenia (Investigations) | 1 (1)
Neutrophil Count Decreased (Investigations) | 1 (1)
Platelet Count Decreased (Investigations) | 1 (2)

LIMITATIONS AND CAVEATS:
After 1 patient was recruited, this trial temporarily closed to allow the first dose of Anti-thymocyte Globulin to be split over two days. Before the modification was written, it was decided to permanently close this study due to competing trials.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No